CLINICAL TRIAL: NCT01353391
Title: Metformin in Women With Type 2 Diabetes in Pregnancy Trial
Acronym: MiTy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOP-106678
Record Dates: First submitted 2011-05-02; First posted 2011-05-13 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; MiTy; Metformin in Women; Type 2 Diabetes Pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Metformin — 500 mg daily OD from randomisation for 2 weeks, then 1000mg BID throughout the duration of pregnancy
  Arms: Metformin
Drug: Placebo Comparator — 500 mg daily OD from randomisation for 2 weeks, then 1000mg BID throughout the duration of pregnancy
  Arms: Placebo

SUMMARY:
Insulin is the standard treatment for the management of type 2 diabetes in pregnancy, however despite treatment with insulin, these women continue to face increased rates of adverse maternal and fetal outcomes. The investigators hypothesize that metformin use, in addition to treatment with insulin, will help with blood sugar control, lower the dose of insulin needed, lower weight gain, and improve baby outcomes.

DETAILED DESCRIPTION:
Type 2 diabetes in pregnancy is increasing in prevalence and these women continue to face increased rates of adverse maternal and fetal outcomes. The investigators hypothesize that metformin use, as an adjunct to insulin, will decrease these adverse outcomes by reducing maternal hyperglycemia, high maternal insulin doses, excessive maternal weight gain and gestational hypertension/pre-eclampsia, all of which should reduce perinatal and neonatal mortality and morbidity. In addition, since metformin crosses the placenta, metformin treatment of the fetus may have a direct beneficial effect on neonatal outcomes. This study is an randomized controlled trial (RCT) that adds metformin to insulin, and is a double-blind, placebo-controlled RCT. The investigators believe that neither metformin alone nor insulin alone will effectively treat this population, and therefore our design, which includes the addition of metformin to insulin, will be the most relevant to our patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are between of 18-45 years of age.
2. (i). Women diagnosed with type 2 diabetes prior to pregnancy, OR (ii). Women with undiagnosed type 2 diabetes diagnosed prior to 20 weeks gestation, defined as women presenting with gestational diabetes before 20 weeks gestation with various combinations, as per Canadian Diabetes Association, including:

   * 2 fasting glucose ≥ 7.0 mmol/L, or
   * 2 HbA1c of ≥0.065 (6.5%) performed in a laboratory using a method that is standardized to the Diabetes Control and Complications Trial (DCCT) assay, or
   * 1 fasting glucose ≥7.0 mmol/L and 1 HbA1c ≥ 0.065 (6.5%) performed in a laboratory using a method that is standardized to the DCCT assay, or
   * 1 fasting glucose ≥ 7.0 mmol/L and 1 two hour (2 hr) ≥ 11.1 on a 75 g Oral Glucose Tolerance Test (OGTT), or
   * 1 HbA1C ≥0.065 (6.5%) performed in a laboratory using a method that is standardized to the DCCT assay and 1 two hour (2 hr) ≥ 11.1 on a 75 g OGTT.
3. Pregnancy gestation between 6+0-22+6 weeks.
4. Live singleton fetus.

Exclusion Criteria:

1. Women who are not on insulin. Women who are on oral hypoglycemic agents will be taken off at the start of the trial and started on insulin prior to randomization.
2. Diabetes diagnosed after 20 weeks gestation.
3. Type 1 diabetes.
4. Known intolerance to metformin.
5. Contraindications to metformin use which include:

(i). Renal insufficiency (defined as serum creatinine of greater than 130 µmol/L or creatinine clearance <60 ml/min) , (ii). Moderate to severe liver dysfunction (defined as liver enzymes (aspartate aminotransferase (AST) and alanine aminotransferase (ALT)) greater than 3 times the upper limit of normal), (iii). Shock or sepsis, and (iv.) Previous hypersensitivity to metformin.

f. Women with significant gastrointestinal problems such as severe vomiting requiring IV fluids or hospitalization, or active Crohn's or colitis.

g. Previous participation in the trial. h. Women who have a fetus with a known potentially lethal anomaly will be excluded. Information regarding congenital anomalies diagnosed after randomization will be recorded.

i. Known higher order pregnancies (twins, triplets, etc). These women will be excluded as they have a higher rate of adverse outcomes and we want to avoid any inequalities if they are unequally distributed between the groups.

j. Presence of acute or chronic metabolic acidosis, including diabetic ketoacidosis.

k. History of diabetic ketoacidosis or history of lactic acidosis. l. Presence of excessive alcohol intake, acute or chronic. m. Presence of congestive heart failure or history of congestive heart failure.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
A composite of: pregnancy loss, preterm birth, birth injury, moderate/severe respiratory distress, neonatal hypoglycemia, and NICU admission > 24 hours. | conception to 28 days after birth

SECONDARY OUTCOMES:
Large for gestational age (LGA) infants | Up to 24 hours after birth
  Defined as greater than the 90th percentile for weight, based on the National canadian fetal growth standards for singleton boys and girls.
Pregnancy loss | Up to 40 weeks gestation
  Spontaneous abortion defined as death of a fetus at <20 weeks gestation; Stillbirth defined as death of a fetus with a birth weight ≥ 500g or at ≥ 20 wks gestational age regardless of birth weight; Neonatal death defined as death of a live born infant within the first 28 days of life or prior to hospital discharge, whichever is later.
Preterm birth | Up to 37 weeks gestation
  Birth < 37 weeks gestation
Respiratory distress | within 72 hours after birth
  Given surfactant via an endotracheal tube and/or requiring assisted positive pressure ventilation within 72 hours after birth.
Neonatal hypoglycemia | NICU admission >24 hours
  A plasma glucose <2.6 mmol/L on one or more occasions, starting at 30-60 minutes after birth, and necessitating intravenous dextrose within the first 48 hours of life.
NICU admission >24 hours | NICU admission >24 hours
  Admission to a neonatal intensive or special care unit for > 24 hours during the initial hospitalization after birth
Cord blood gases pH <7.0 | Within 4 hours of birth
Hyperinsulinemia as measured by elevated cord blood C-peptide | Within 4 hours of birth
  A cord serum C-peptide value > 1.7 ug/L (which is >90th percentile of values for the total cohort of participants in the HAPO trial) will be defined as hyperinsulinemia.
Maternal glycemic control as measured by HbA1c and capillary glucose measurements. | Up to 40 weeks gestation
  Gestational age at testing will be recorded. All downloaded glucose results will be transmitted on a regular basis to a central site for future analysis. Monthly correlations will be done with the laboratory during routine monthly blood draws.
Maternal hypoglycemia | Up to 40 weeks gestation
  Maternal hypoglycemia defined as mild (<3.6, symptomatic and asymptomatic or requiring treatment), or severe (loss of consciousness or confusion requiring assistance) will be documented at each visit.
Maternal weight gain | Up to 40 weeks gestation
  The first and last weight will be obtained at the first and last visit in pregnancy, whether they be done by the endocrinologist, family physician or obstetrician.
Maternal insulin doses | Up to 40 weeks gestation
  Maternal insulin doses (overall amount and number of patients that are taking 'high' insulin doses defined as 2 Units/kg or more per day)
Pre-eclampsia, and/or gestational hypertension | Up to 40 weeks gestation
  Gestational hypertension: New onset of hypertension in pregnancy ≥ 20 weeks gestation in a woman with previously normal blood pressure, defined as diastolic blood pressure of ≥ 90 mmHg, taken on 2 occasions or placed on antihypertensive medication and without proteinuria.
  Pre-eclampsia: please refer to protocol for definition
Sepsis | Up to 28 days after birth
  A positive blood and/or cerebral spinal fluid culture during the neonatal hospital stay.
Hyperbilirubinemia | First 7 days of life
  Significant jaundice was present based on bilirubin levels requiring treatment with phototherapy> 6 continuous hours, or an exchange transfusion, or receiving intravenous gamma globulin, or requiring readmission into hospital during the first 7 days of life.
Number of hospitalizations | Up to 40 weeks gestation
  Number of hospitalizations prior to admission for delivery and the duration of hospital stays for the mother prior to admission for delivery and associated with delivery.
Rate of caesarean-section | Up to 40 weeks gestation
Duration of hospital stay for infant. | Up to 28 days after birth
  Duration of hospital stay for infant associated with his/her birth until the first discharge home
Fetal fat mass | Up to 7 days after birth
  Fetal fat mass compared with women treated with insulin plus placebo
Birth Injury | Up to 7 days after birth
  Defined as any of the following: spinal cord injury, basal skull fracture or depressed skull fracture, clavicular fracture, long bone fracture, subdural or intracerebral hemorrhage or any kind
Shoulder dystocia | At delivery
  Documentation of any shoulder dystocia in the delivery records, plus 3 or more of the following: McRoberts maneuver, suprapubic maneuver, episiotomy, delivery of the posterior arm, Woods maneuver, Rubins maneuver, All fours Gaskins maneuver, intentional fracture of the clavicle, and/or Zavenelli maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Denice Feig, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- The Centre for Mother, Infant, and Child Research, Sunnybrook Research Institute, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Feig DS, Donovan LE, Zinman B, Sanchez JJ, Asztalos E, Ryan EA, Fantus IG, Hutton E, Armson AB, Lipscombe LL, Simmons D, Barrett JFR, Karanicolas PJ, Tobin S, McIntyre HD, Tian SY, Tomlinson G, Murphy KE; MiTy Collaborative Group. Metformin in women with type 2 diabetes in pregnancy (MiTy): a multicentre, international, randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2020 Oct;8(10):834-844. doi: 10.1016/S2213-8587(20)30310-7. PMID 32946820
- [Derived] Feig DS, Murphy K, Asztalos E, Tomlinson G, Sanchez J, Zinman B, Ohlsson A, Ryan EA, Fantus IG, Armson AB, Lipscombe LL, Barrett JF; MiTy Collaborative Group. Metformin in women with type 2 diabetes in pregnancy (MiTy): a multi-center randomized controlled trial. BMC Pregnancy Childbirth. 2016 Jul 19;16(1):173. doi: 10.1186/s12884-016-0954-4. PMID 27435163